CLINICAL TRIAL: NCT04076553
Title: Augmenting Cognitive Behavioral Therapy for Binge Eating Disorder and Bulimia Nervosa With Inhibitory Control Training
Brief Title: Augmenting Cognitive Behavioral Therapy With Inhibitory Control Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1904007136
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Binge-Eating Disorder; Bulimia Nervosa
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the ICT or ICT sham condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators, therapists, and graduate student assessors will be blinded to treatment condition. The only staff member who cannot be blinded to condition is the study coordinator; she will be aware of condition because of managing randomization and assisting participants in the downloading of the intervention to participants' computers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT + ICT (Active Comparator): Participants randomized to the ICT condition will complete a computerized ICT training at home during the first 4 weeks of treatment and ICT "boosters" following their treatment sessions during weeks 5-12.
  Interventions: Behavioral: CBT; Behavioral: ICT
- CBT + sham (Sham Comparator): Participants randomized to the sham condition will complete a computerized sham ICT training at home during the first 4 weeks of treatment and sham ICT "boosters" following their treatment sessions during weeks 5-12. The shame will contain the same proportion of food as non-food but no inhibitory training component.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — Participants will complete 12 sessions of CBT
Behavioral: ICT — Participants will complete 4 weeks of daily inhibitory control trainings and "booster" ICT trainings following CBT treatment in weeks 5-12
  Arms: CBT + ICT

SUMMARY:
The primary aim of this study is to determine whether a computerized inhibitory control training (ICT) will improve CBT treatment outcomes for Bulimia Nervosa and Binge Eating Disorder.

DETAILED DESCRIPTION:
This study involves a brief phone screen and baseline assessment to determine eligibility. Participants who are eligible for the study will receive 12 sessions of CBT treatment and will be randomly assigned to an ICT or ICT sham condition which will consist of completing ICT computer tasks on a daily basis during the first four weeks of treatment and booster sessions following treatment. Participants will also complete research assessments at mid-treatment, post-treatment, and 3-month follow-up intervals. Research assessments include a battery of questionnaires, computerized tasks, interviews, and behavioral tasks.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* meet DSM-5 criteria for Bulimia Nervosa (i.e., at least one episode of binge eating and compensatory behavior per week on average for the past 3 months) or Binge Eating Disorder (i.e., at least one episode of binge eating per week on average for the past 3 months).
* be stable on psychiatric medications for at least 3 months

Exclusion Criteria:

* have a diagnosis of anorexia nervosa or a BMI < 18.5
* have extreme malnutrition or other medical complications that require acute hospitalization
* are at acute suicide risk
* are currently experiencing other severe psychopathology that would require a more intensive or specialized treatment program than the current study provides (e.g. severe depression, active psychotic disorder)
* have previously completed a trial of CBT for Bulimia Nervosa or Binge Eating Disorder
* have a diagnosis of an intellectual disability or autism spectrum disorder
* currently taking stimulant medications
* score of 95% or higher on 550ms block of Go/No-Go assessment task, indicating high inhibitory control at Baseline

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination (EDE) | Change in binge frequency from baseline to post-treatment and 3-month follow-up
  The Eating Disorder Examination is a widely utilized, semi-structured interview for the assessment of eating disorder symptoms and the binge-eating module will be used to determine binge episode frequency.

SECONDARY OUTCOMES:
Food Frequency Questionnaire (FFQ) | Change from baseline to post-treatment and 3-month follow up
  A modified version of the Food Frequency Questionnaire will be used to examine changes in binge eating on specific foods in the last month

OTHER OUTCOMES:
Go/No-Go (GNG) | Change from baseline to post-treatment and 3-month follow up
  Performance on the Go/No-Go computer task will be used to assess changes in inhibitory control
Laboratory Sham Taste Test | Change from baseline to post-treatment and 3-month follow up
  An ecologically valid measure of inhibitory control specific to eating behavior, this task measures the amount of food that a participant consumes during a 10min interval when asked to taste the food presented

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Manasse, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Butler RM, Lampe E, Trainor C, Manasse SM. Fear of weight gain during cognitive behavioral therapy for binge-spectrum eating disorders. Eat Weight Disord. 2023 Mar 6;28(1):29. doi: 10.1007/s40519-023-01541-8. PMID 36879078